CLINICAL TRIAL: NCT03869996
Title: Randomised Controlled Study Comparing Fast Track and Standard Care Protocol on the Functional Outcomes and Hospital Stay of Total Knee Arthroplasty
Brief Title: Total Knee Arthroplasty: Fast Track Protocol is the Future?
Acronym: FastTrack-G
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0001094
Record Dates: First submitted 2019-02-14; First posted 2019-03-11 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis, Knee; Arthropathy of Knee
Keywords: fast track care; total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fast track total knee arthroplasties (Active Comparator): patients treated using fast track care protocol
  Interventions: Procedure: fast track care protocol
- standard care total knee arthroplasties (Active Comparator): patients treated using standard care protocol
  Interventions: Procedure: standard care protocol

INTERVENTIONS:
Procedure: fast track care protocol — fast track care consists in educational preoperative preparation for patients, particular strategies for controlling pain and bleeding and intensive early rehabilitation protocol.
  Arms: fast track total knee arthroplasties
Procedure: standard care protocol — standard care protocol consists in the same surgical intervention without educational preoperative preparation for patients and intensive early rehabilitation protocol.
  Arms: standard care total knee arthroplasties

SUMMARY:
Fast-track total knee arthroplasty (TKA) is a well-established concept including optimized logistics and evidence-based treatment, focusing on minimizing surgical stress and improved post-operative recovery. The aim of this protocol is to compare the standard care and fast track total knee arthroplasties in terms of functional and subjective outcomes, hospital staying, number of transfusions and analgesic consumption.

DETAILED DESCRIPTION:
The aim of this protocol is to compare standard care and fast track total knee arthroplasties. The fast track care consists of:

* preoperative educational lesson in which orthopedic surgeon, anesthesiologist and physiotherapist illustrate the operative and post operative path to the patients
* antalgic protocol administered only orally
* early rehabilitation care. The day of the surgical operation, the physiotherapist helps the patient reach the upright position.

The standard care consists of usual antalgic and physiotherapy post-operative care:

* Antalgic protocol consist in intravenous drugs
* the first physiotherapy session is the day after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by knee osteoarthritis, eligible for primary total knee arthroplasty
* BMI < 32
* Time up ang go test </= 12 seconds
* American Society of Anesthesiologists physical status classification system (ASA) </= 2
* preoperative hemoglobin (HB) >13 g/dl
* patients eligible for spinal anesthesia
* presence of a care-giver

Exclusion Criteria:

* psychiatric diseases
* preoperative use of crutches
* ASA > 3
* preoperative HB < 13 g/dl

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Early functional outcomes | Third post operative day
  Early functional outcomes are collecting using Lowa Level of Assistance(ILOA) during the third post-operative day. This scale is able to provide data on the autonomy reached by the patient in the first postoperative period going to investigate five main motor activities (get up from supine to seated, from sitting to standing position, walk around, take three steps, the speed of walking). the total score can vary from 0 to 50, where 50 indicates better functional results.

SECONDARY OUTCOMES:
hospital staying | Third day after surgery
  The collection of hospital stay for each patient. The fast track expecting hospital stay is three days.
Incidence of early major complications | Third day after surgery
  The collection of acute infection and early fracture
Number of transfusions | Third day after surgery
  the collection of number of transfusions during hospital staying
Analgesic consumption | Third day after surgery
  The request for analgesic rescue in relation to fast track standard analgesic scheme
Knee Society Score (KSS) at 6 weeks | 6 weeks after surgery
  The collection of functional outcomes score KSS at 6 weeks. The Knee Society Score (KSS) is mixed outcome measure that's both objective (physician input) and subjective (patient input). A score between 80 and 100 is considered excellent, between 70 and 79 is considered good, between 60 and 69 is considered fair and below 60 is considered poor.
Knee Society Score (KSS) at third month | third month after surgery
  The collection of functional outcomes score KSS at third month. The Knee Society Score (KSS) is mixed outcome measure that's both objective (physician input) and subjective (patient input). A score between 80 and 100 is considered excellent, between 70 and 79 is considered good, between 60 and 69 is considered fair and below 60 is considered poor.
Knee Society Score (KSS) at sixth month | sixth month after surgery
  The collection of functional outcomes score KSS at sixth month. The Knee Society Score (KSS) is mixed outcome measure that's both objective (physician input) and subjective (patient input). A score between 80 and 100 is considered excellent, between 70 and 79 is considered good, between 60 and 69 is considered fair and below 60 is considered poor.
Knee Society Score (KSS) at twelfth month | twelfth month after surgery
  The collection of functional outcomes score KSS at twelfth month. The Knee Society Score (KSS) is mixed outcome measure that's both objective (physician input) and subjective (patient input). A score between 80 and 100 is considered excellent, between 70 and 79 is considered good, between 60 and 69 is considered fair and below 60 is considered poor.
Oxford Score (OS) at 6 weeks | 6 weeks after surgery
  The collection of functional outcomes score OS at 6 weeks. The Oxford Score is a 12-item patient-reported outcomes (PRO) specifically designed and developed to assess function and pain after total knee replacement surgery. Each question is scored from 0 to 4 (0 being the worst outcome and 4 being the best). The overall score is the sum of all items and can range from 0 to 48, with higher scores corresponding to better outcomes.
Oxford Score (OS) at third month | third month after surgery
  The collection of functional outcomes score OS at third month. The Oxford Score is a 12-item patient-reported outcomes (PRO) specifically designed and developed to assess function and pain after total knee replacement surgery. Each question is scored from 0 to 4 (0 being the worst outcome and 4 being the best). The overall score is the sum of all items and can range from 0 to 48, with higher scores corresponding to better outcomes.
Oxford Score (OS) at sixth month | sixth month after surgery
  The collection of functional outcomes score OS at sixth month. The Oxford Score is a 12-item patient-reported outcomes (PRO) specifically designed and developed to assess function and pain after total knee replacement surgery. Each question is scored from 0 to 4 (0 being the worst outcome and 4 being the best). The overall score is the sum of all items and can range from 0 to 48, with higher scores corresponding to better outcomes.
Oxford Score (OS) at twelfth month | twelfth month after surgery
  The collection of functional outcomes score OS at twelfth month. The Oxford Score is a 12-item patient-reported outcomes (PRO) specifically designed and developed to assess function and pain after total knee replacement surgery. Each question is scored from 0 to 4 (0 being the worst outcome and 4 being the best). The overall score is the sum of all items and can range from 0 to 48, with higher scores corresponding to better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Stagni, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided